CLINICAL TRIAL: NCT01152632
Title: Acupuncture Treatment for Migraine: a Functional Magnetic Resonance Imaging Study
Brief Title: Acupuncture for Migraine: a Functional Magnetic Resonance Imaging (fMRI) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 30930112/C190301
Record Dates: First submitted 2010-06-27; First posted 2010-06-29 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2012-08

CONDITIONS: Migraine
Keywords: acupuncture; migraine; specific acupoints; brain network
MeSH Terms: conditions — Migraine Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- specific points of Bladder meridian and Shanjiao meridian (Experimental): In traditional Chinese acupuncture theory, Bladder meridian and Shanjiao meridian have been considered as the main pathological meridian location of migraine. Meanwhile, specific points on both meridians have been used widely in its treatment for a long time.
  Interventions: Other: manual acupuncture
- non-specific points of Bladder meridian and Shanjiao meridian (Experimental): Non-specific points of Shaoyang meridians are also used in cure of migraine. It is conventionally thought to be less effective using non-specific points than specific ones.
  Interventions: Other: manual acupuncture
- specific points of Stomach meridian (Active Comparator): Specific points of Stomache meridian for migraine were searched in Chinese ancient data. And this group is set to compare with specific points of Shaoyang meridians for their possible different brain networks.
  Interventions: Other: manual acupuncture
- non-acupoints (Placebo Comparator): Three non-acupoints were chosen,two of which were located on the arm and one one the leg.
  Interventions: Other: manual acupuncture
- waiting list (No Intervention)

INTERVENTIONS:
Other: manual acupuncture — thirty minutes duration every time, five times per week for one course, a total four courses
  Other Names: acupuncture
  Arms: non-acupoints; non-specific points of Bladder meridian and Shanjiao meridian; specific points of Bladder meridian and Shanjiao meridian; specific points of Stomach meridian

SUMMARY:
Selecting acupoints along meridians is the predominant principle in acupuncture treatment, and it is also considered to ensure acupuncture efficacy. This experiment is to investigate whether specific brain networks gradually come in formation in accordance with this kind of acupoint selection methods.

DETAILED DESCRIPTION:
Every participants in the four intervention groups will go through functional magnetic imaging (fMRI) scan four times: the 1st scan will be performed at their baselines; the 2nd scan will be done after 2 courses (10 times) acupuncture treatment; the 3rd scan will be performed when the 4 courses end; the 4th scan will be operated after three-month enrollment.

Volunteers in waiting list group will undergo the above scans at the same time points in exception of acupuncture treatment.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of non-aura Migraine formulated by the international headache society in 2004

Exclusion Criteria:

* people with other types of headache
* people with organic cerebral disorders
* people with primary disorders
* people in moderate or severe anxiety or depression
* people in pregnancy

Ages: 17 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
improvement of headache frequency | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fanrong Liang, Master, Study Chair — Chengdu University of Traditional Chinese Medicine
Locations (1):
- Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Li Z, Zhou J, Lan L, Cheng S, Sun R, Gong Q, Wintermark M, Zeng F, Liang F. Concurrent brain structural and functional alterations in patients with migraine without aura: an fMRI study. J Headache Pain. 2020 Dec 7;21(1):141. doi: 10.1186/s10194-020-01203-5. PMID 33287704